CLINICAL TRIAL: NCT02745353
Title: A Phase II, Randomized, Single Center, Pilot Feasibility Study to Evaluate Naloxegol for Opioid-Induced Constipation in Cancer Patients
Brief Title: Naloxegol in Cancer Opioid-Induced Constipation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Couldn't enough accrue patients
Sponsor: Joseph Ma (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Joseph Ma, Associate Clinical Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 160121
Record Dates: First submitted 2016-04-15; First posted 2016-04-20 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Constipation
Keywords: Cancer; Constipation; Opioid
MeSH Terms: conditions — Constipation; Neoplasms | interventions — naloxegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Patients in Arm A will receive a single daily dose of 25mg naloxegol for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover treatment period in which the patient will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication.
  Interventions: Drug: naloxegol
- B (Active Comparator): Patients in Arm B will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover period in which the patient will receive a single daily dose of 25mg naloxegol.
  Interventions: Drug: naloxegol

INTERVENTIONS:
Drug: naloxegol
  Other Names: MOVANTIK

SUMMARY:
The purpose of this study is to compare the effect of naloxegol versus the patient's usual care in treating opioid-induced constipation, as well as the effect on the patient's quality of life and how much pain is experienced. Also, the purpose of this study is to compare whether treatment with naloxegol versus usual care has any impact on the number of hospital or clinic visits or telephone calls to the patient's physician that are related to constipation, and to determine the patient's preference for continuing to receive naloxegol as treatment for opioid-induced constipation.

DETAILED DESCRIPTION:
Opioid-induced constipation (OIC) is a common symptom in patients with cancer-related pain and requires burdensome self-titration of laxatives for prophylaxis and treatment. Consequently, naloxegol may have an important role in this setting. Naloxegol has been evaluated in relieving OIC with cancer patients in a randomized, double blind, placebo-controlled trial over 4 weeks with a 12-week extension phase. However, accrual was challenging and the trial was closed early. Given the complexity of cancer and its treatment, a key first step is to determine if evaluating naloxegol versus standard of care is feasible in the management of OIC in this setting.

Subjects will receive naloxegol 25mg daily or usual care for a 2-week initial treatment period followed by 3-day washout period, then a 2-week crossover treatment period where subjects will receive naloxegol or usual care. Treatment assignment during the initial and crossover treatment periods will be dictated by the randomization arm. Subjects will also have the option to participate in a 12-week extension phase of naloxegol.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to 18 years old.
* Eastern Cooperative Oncology Group (ECOG) less than or equal to 3.
* Glomerular filtration rate (GFR) greater than or equal to 30 ml/min/1.73m2 by Modification of Diet in Renal Disease (MDRD).
* Corrected serum calcium level less than or equal to 10.5 mg/dL.
* Estimated life expectancy greater than or equal to 6 months.
* Negative pregnancy test prior to initiating study treatment for females of childbearing potential.

Exclusion Criteria:

* Patients receiving the following medications within 3 days of Study Day 1 and/or are planned to receive throughout the duration of the study period: opioid antagonist, mixed antagonist, a strong CYP3A4 and/or P-glycoprotein (P-gp) inhibitor, a moderate CYP3A4 and/or P-gp inhibitor, and/or a strong CYP3A4 inducer.
* Concurrent total parenteral nutrition and/or use of metoclopramide.
* Patients at high risk for bowel perforation.
* Constipation that was not primarily caused by opioids in the investigator's medical opinion.
* A condition that may have affected the permeability of the blood-brain barrier (e.g., known brain metastases, meningeal metastases, brain injury, multiple sclerosis, recent brain injury, uncontrolled epilepsy)
* Patient has clinically active diverticular disease.
* Past medical history of irritable bowel syndrome, signs of active gastrointestinal (GI) bleeding, acute surgical abdomen, bowel stents, indwelling peritoneal catheter, mechanical GI obstruction, fecal impaction, or fecal ostomy.
* Patient has motility/neurologic disorders including autonomic failure (spinal cord lesions, tumor invasion of nerves) and/or poorly controlled endocrine/metabolic disorders (hypercalcemia, hypokalemia, diabetes, hypothyroidism), as determined by the investigator.
* Uncontrolled cancer pain despite analgesic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06-22 (Actual); Study Completion 2017-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ma, PharmD, Principal Investigator — UCSD
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- A- Naloxegol/ Standard of Care: Patients in Arm A will receive a single daily dose of 25mg naloxegol for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover treatment period in which the patient will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication.
  naloxegol
- B- Standard of Care/ Naloxegol: Patients in Arm B will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover period in which the patient will receive a single daily dose of 25mg naloxegol.
  naloxegol
Period: First Intervention (2 Weeks)
Arm/Group | A- Naloxegol/ Standard of Care | B- Standard of Care/ Naloxegol
Started | 4 | 3
Completed | 1 | 1
Not Completed | 3 | 2
Period: Washout (3 Days)
Arm/Group | A- Naloxegol/ Standard of Care | B- Standard of Care/ Naloxegol
Started | 1 | 1
Completed | 1 | 1
Not Completed | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | A- Naloxegol/ Standard of Care | B- Standard of Care/ Naloxegol
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- A- Naloxegol/Standard of Care: Patients in Arm A will receive a single daily dose of 25mg naloxegol for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover treatment period in which the patient will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication.
  naloxegol
- B - Standard of Care/Naloxegol: Patients in Arm B will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover period in which the patient will receive a single daily dose of 25mg naloxegol.
  naloxegol
- Total: Total of all reporting groups
Arm/Group | A- Naloxegol/Standard of Care | B - Standard of Care/Naloxegol | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completed Naloxegol 25mg and the Number of Participants That Completed Standard of Care
Description: completion of treatment defined as participants receiving all single daily doses for 2 weeks
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Arm A (Naloxegol/Standard of Care): Patients in Arm A will receive a single daily dose of 25mg naloxegol for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover treatment period in which the patient will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication.
  naloxegol
- Arm B (Standard of Care/ Naloxego): Patients in Arm B will receive the treating physician's usual care for OIC using a stimulant laxative + rescue medication for the 2-week initial treatment period, followed by a 3-day washout period and 2-week crossover period in which the patient will receive a single daily dose of 25mg naloxegol.
  naloxegol
Arm/Group | Arm A (Naloxegol/Standard of Care) | Arm B (Standard of Care/ Naloxego)
Number analyzed (Participants) | 4 | 3
Participants
  Naloxegol | 4 | 3
  Standard of Care | 1 | 1

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Naloxegol: All patients who received a single daily dose of 25 mg Naloxegol during the entire study duration
- Standard of Care: All patients who received Standard of Care during the entire study duration
Arm/Group | Naloxegol | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/5 | 1/4
Other Adverse Events (participants affected / at risk) | 3/5 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naloxegol (N=5) | Standard of Care (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Fever (Immune system disorders) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 2 (3) | 1 (1)
platelet count decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naloxegol (N=5) | Standard of Care (N=4)
Hypoalbuminemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT02745353/Prot_SAP_000.pdf